CLINICAL TRIAL: NCT07276841
Title: Digital Occlusal Analysis and Bite Force Evaluation of Pulp Treated Primary Molars Restored With Zirconia Crowns Using T-Scan: An Experimental Before-and-After Study
Brief Title: Digital Occlusal Analysis and Bite Force Evaluation of Primary Molars Restored With Zirconia Crowns Using T-Scan
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Lama Hatem Mohamed Kamal Belal, Master's Student, Department of Pediatric Dentistry, Cairo University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PEDS-TSCAN-ZC-2025-01
Record Dates: First submitted 2025-11-30; First posted 2025-12-11 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-11

CONDITIONS: Dental Occlusion; Primary Teeth; Pulp-treated Primary Molars; Zirconia Crowns
Keywords: Occlusion; Bite Force; Pediatric Dentistry; Zirconia Crown; T-Scan; Primary Teeth; Restorative Dentistry
MeSH Terms: conditions — Bites and Stings

STUDY DESIGN:
Intervention Model Description: This is a single-group, before-and-after interventional study. All participants will receive the intervention, which is restoration of pulp-treated primary molars with prefabricated zirconia crowns. Outcome measures, including bite force and occlusal adaptation, will be recorded prior to crown placement (baseline) and at follow-up visits 2 weeks and 4 weeks post-restoration to assess functional adaptation over time.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Zirconia Crown Restoration of Pulp-Treated Primary Molars (Experimental): All participants will receive pulp therapy and restoration of primary molars with prefabricated zirconia crowns. Bite force and occlusal contacts will be measured using the T-Scan digital occlusal analysis system at baseline, 2 weeks, and 4 weeks post-restoration. Participants act as their own control, with pre-restoration measurements compared to post-restoration outcomes. No comparison or additional study arms are included.
  Interventions: Procedure: Pulp Therapy and Zirconia Crown Restoration of Primary Molars with T-Scan Occlusal Analysis

INTERVENTIONS:
Procedure: Pulp Therapy and Zirconia Crown Restoration of Primary Molars with T-Scan Occlusal Analysis — Participants will receive pulp therapy followed by restoration of primary molars with prefabricated zirconia crowns according to standard pediatric dental protocols. Occlusal function and bite force will be assessed using the T-Scan digital occlusal analysis system at baseline, and at 2 and 4 weeks post-restoration. This intervention combines a therapeutic dental procedure with objective, instrumented measurement of occlusal adaptation, allowing participants to act as their own controls. Follow-up visits will monitor crown fit, occlusal contacts, and bite force changes over time.

SUMMARY:
The goal of this observational study is to evaluate the adaptation of occlusion and bite force after zirconia crown restoration in children with pulp-treated primary molars. The main questions it aims to answer are:

How does occlusion adapt after placement of zirconia crowns?

Does bite force change following crown restoration?

Participants will:

Undergo routine pulp treatment and restoration of primary molars with zirconia crowns.

Have bite force and occlusal contacts measured using the T-Scan digital occlusal analysis system before and after crown placement.

DETAILED DESCRIPTION:
his observational before-and-after study is designed to evaluate occlusal adaptation and functional outcomes in children undergoing pulp treatment and restoration of primary molars with zirconia crowns. The study employs the T-Scan Novus digital occlusal analysis system to objectively measure bite force distribution and occlusal contact patterns.

After informed consent is obtained from parents or legal guardians, baseline occlusal measurements will be collected using the T-Scan system prior to crown placement. Standard pulp therapy and restoration procedures will be performed according to pediatric dental protocols. Prefabricated zirconia crowns will be selected and fitted, with occlusal adjustments performed as needed to ensure proper seating and contact.

Participants will be scheduled for follow-up visits at 2 weeks and 4 weeks post-restoration, during which occlusal measurements will be repeated using the T-Scan system. These follow-ups are designed to track the progressive adaptation of occlusion and detect any functional changes following crown placement.

Additional technical considerations include:

Calibration of the T-Scan system prior to each measurement session.

Standardized patient positioning during measurements to ensure reproducibility.

Recording of bite force in a controlled environment, minimizing variables such as head posture and tongue position.

Monitoring of crown integrity and fit during follow-up visits.

This study will provide detailed insight into the functional adaptation of primary molars after zirconia crown restoration, including occlusal contact patterns and bite force distribution, contributing to evidence-based recommendations for pediatric restorative dentistry.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 6 to 9 years.
* Both boys and girls can participate.
* A pulp-treated primary molar (pulpotomy) that is healthy and shows no pain, no swelling, no mobility, and no radiographic problems (such as internal resorption or infection).
* The lower first permanent molar must be erupted.
* The child is cooperative during dental treatment (positive behavior on the Frankl scale).
* The child has no missing teeth.
* The child has a normal bite (normal overjet and overbite).
* The child is generally healthy with no systemic diseases, to ensure they can attend follow-ups.

Exclusion Criteria:

* Children with medical conditions or who are uncooperative during dental care.
* Children with parafunctional habits, such as teeth grinding (bruxism), thumb-sucking, or other habits that may affect bite-force measurements.
* Teeth that are close to falling out, have severe root resorption, or need extraction.
* Teeth with deep cavities below the gum line that prevent proper crown placement.
* Teeth that are mobile (Miller's Grade 2 or higher).
* Teeth that have had previous pulp therapy other than the included pulpotomy.
* Children who are unable to attend follow-up visits or whose parents do not agree to participate.

Ages: 6 Years to 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 11 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Mean Bite Force | Baseline (pre-operative), immediate post-operative, 2 weeks post-operative, 4 weeks post-operative
  Bite force will be measured using the T-Scan digital occlusal analysis system. Participants will bite on the sensor in a standardized position, and the system will record bite force as a percentage of total occlusal force distributed among teeth. This measure reflects functional adaptation of occlusion after crown placement.

SECONDARY OUTCOMES:
Vertical Dimension | Baseline (pre-operative), immediate post-operative, 2 weeks post-operative, 4 weeks post-operative
  Vertical dimension will be measured using a digital vernier caliper. Before local anesthesia, the vertical distance (overbite) at the cuspid will be measured, with the child seated upright in maximum intercuspal position. The most prominent incisal edge of the maxillary cuspid will be marked, and the vertical distance to the mandibular cuspid measured. Measurements will be recorded at pre-operative, immediate post-operative, and 1, 2, and 4 weeks post-operative to assess changes in occlusion following operative zirconia crown placement.
Parental Rating of Esthetic Satisfaction | immediate post-operative and 4 weeks post-operative
  Description: Parents will rate the appearance of the treated teeth using a 5-point Likert scale (1 = very dissatisfied, 5 = very satisfied). This measure assesses parental satisfaction with the esthetics of the operative zirconia crown placement at each follow-up
Parental Rating of Treatment Impact on Child | immediate post-operative and 4 weeks post-operative
  Parents will complete a structured questionnaire assessing the perceived impact of zirconia crown placement on their child's oral health, appearance, and psychosocial comfort. The questionnaire consists of 5 items, each scored on a 5-point Likert scale, where:
  1 = Not at all satisfied
  5 = Very much satisfied
  Items include:
  Oral health of the child improved after crowns
  Parents' concern about appearance before the crowns
  Child avoided smiling before the crowns
  Child smiled after crowns
  Crowns improved the appearance of the child's teeth
  Higher scores indicate greater positive impact of the treatment on the child's oral health and well-being

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry, Cairo University, Cairo, Giza Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Umapathy Thimmegowda and Radhakrishnan, A. (2023). Application of Tekscan in Pediatric Dentistry: A Review. Researchgate, pp.132-142. doi:https://doi.org/10.9734/bpi/cidhr/v1/6603a.
- [Background] Nair K, Chikkanarasaiah N, Poovani S, Thumati P. Digital occlusal analysis of vertical dimension and maximum intercuspal position after placement of stainless steel crown using hall technique in children. Int J Paediatr Dent. 2020 Nov;30(6):805-815. doi: 10.1111/ipd.12647. Epub 2020 May 7. PMID 32248585
- [Background] Panwar, M., Gupta, S., Singh, U., Das, A., & Isha, S. (2023). Role of Intraoral Scanners in Pediatric Dentistry. International Journal of Medical and Dental Sciences, 2071-2076. https://doi.org/10.18311/ijmds/2023/646
- [Background] Rahate I, Fulzele P, Thosar N. Comparative evaluation of clinical performance, child and parental satisfaction of Bioflx, zirconia and stainless steel crowns in pediatric patients. F1000Res. 2023 Dec 21;12:756. doi: 10.12688/f1000research.133464.2. eCollection 2023. PMID 38911945
- [Background] Haghgoo R, Abbasi F. Clinical and Radiographic Success of Pulpotomy with MTA in Primary Molars: 30 Months Follow up. Iran Endod J. 2010 Fall;5(4):157-60. Epub 2010 Nov 15. PMID 23130045
- [Background] Sowmya Gujjar Vishnurao, Madhusudan Astekar and Aggarwal, A. (2023). T scan - A review on an occlusal indicator in dentistry. International Journal of Maxillofacial Imaging, 9(3), pp.119-124. doi:https://doi.org/10.18231/j.ijmi.2023.021
- [Background] Abutayyem H, M Annamma L, Desai VB, Alam MK. Evaluation of occlusal bite force distribution by T-Scan in orthodontic patients with different occlusal characteristics: a cross sectional-observational study. BMC Oral Health. 2023 Nov 20;23(1):888. doi: 10.1186/s12903-023-03544-4. PMID 37986159
- [Background] Alzanbaqi SD, Alogaiel RM, Alasmari MA, Al Essa AM, Khogeer LN, Alanazi BS, Hawsah ES, Shaikh AM, Ibrahim MS. Zirconia Crowns for Primary Teeth: A Systematic Review and Meta-Analyses. Int J Environ Res Public Health. 2022 Feb 28;19(5):2838. doi: 10.3390/ijerph19052838. PMID 35270531
- [Result] Maheshkumar K, Chowdhary N, Chowdharry R, Vundela RR, Sonnahalli NK, Anuraaga AT. Bite force evaluation at maximal intercuspal position: An in vivo comparative study between stainless steel and zirconia crowns on primary molar teeth. J Indian Soc Pedod Prev Dent. 2023 Apr-Jun;41(2):89-97. doi: 10.4103/jisppd.jisppd_156_23. PMID 37635466
- [Result] Bozhkova TP. The T-SCAN System in Evaluating Occlusal Contacts. Folia Med (Plovdiv). 2016 Apr-Jun;58(2):122-30. doi: 10.1515/folmed-2016-0015. PMID 27552789